CLINICAL TRIAL: NCT05873036
Title: Comparison of Aerobic Training and Progressive Resistance Training to Improve Functional Ability After Breast Cancer Surgery
Brief Title: Comparison of AT & PR Training to Improve Functional Ability After Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/547
Record Dates: First submitted 2023-03-18; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Training (Other)
  Interventions: Diagnostic Test: Aerobic Training
- Progressive Resistance Training (Experimental)
  Interventions: Diagnostic Test: Progressive Resistance Training

INTERVENTIONS:
Diagnostic Test: Aerobic Training — Aerobic Training to Improve Functional Ability After Breast Cancer Surgery
  Arms: Aerobic Training
Diagnostic Test: Progressive Resistance Training — Progressive Resistance Training to Improve Functional Ability After Breast Cancer Surgery
  Arms: Progressive Resistance Training

SUMMARY:
To determine the effect of aerobic training and progressive resistance training to improve upper limb functional ability after breast cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* a) Breast cancer female survivors eligible under 35-65 years complaining of cancer-related fatigue.

  b) Adjunctive radiotherapy or underwent surgery (lumpectomy or mastectomy), willing to participate will be included in the study.

  c) Shoulder pain d) Decreased ROM e) Primary unilateral BC, ALND, no distant metastases, no previous ALND on the contra lateral side f) No previous history of arm lymph edema

Exclusion Criteria:

- a) Survivors with other concurrent metastasis anywhere else in the body, diagnosed case of any cardiac or respiratory condition, contra-indicated for exercise training (severe dyspnea, chest pain, severe nausea, ataxia, dizziness etc.) b) Any other neurological or recent musculoskeletal problems were excluded from the study.

c) Bilateral mastectomy d) Adjunctive chemotherapy

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale (NPRS) | 6 Months
Goniometer Tool | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudhary Muhammad Akram Teaching and research hospital, Jinnah Hospital Lahore and Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No